CLINICAL TRIAL: NCT04902599
Title: Renuvion/J-Plasma for Subdermal Skin Tightening and Contouring of the Upper Arms: a Randomized, Intra-patient, Left-right Arm, Non-inferiority Clinical Trial Comparing Vaser to Blunt Dissection for Site Preparation.
Brief Title: Renuvion/J-Plasma for Subdermal Skin Tightening and Contouring of the Upper Arms: Dissection Technique Comparison
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Dr. Smart is leaving the instution.
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Smart, Assistant Professor, Dermatology, Principal Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB_00127330
Record Dates: First submitted 2021-04-28; First posted 2021-05-26 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Subdermal Skin Tightening

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Technique Comparison Trial
Who Masked: Outcomes Assessor
Masking Description: A blinded assessor will review the results to determine if there is a significant difference in the two techniques by looking at the photos once the study is over.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaser ulstrasound-assisted dissection technique (Active Comparator): Patient's arm that undergoes treatment using Renuvion/j-Plasma for subdermal skin tightening and contouring with the Vaser ultrasound-assisted dissection technique.
  Interventions: Procedure: Renuvion/j-Plasma procedure using ultrasound-guided dissection technique
- Blunt dissection technique (Active Comparator): Patient's arm that undergoes treatment using Renuvion/j-Plasma for subdermal skin tightening and contouring with blunt dissection technique.
  Interventions: Procedure: Renuvion/j-Plasma procedure using blunt dissection technique

INTERVENTIONS:
Procedure: Renuvion/j-Plasma procedure using blunt dissection technique — Renuvion/j-Plasma procedure using blunt dissection technique
  Arms: Blunt dissection technique
Procedure: Renuvion/j-Plasma procedure using ultrasound-guided dissection technique — Renuvion/j-Plasma procedure using ultrasound-guided dissection technique.
  Arms: Vaser ulstrasound-assisted dissection technique

SUMMARY:
The Renuvion/J-plasma cold atmospheric plasma device has been in clinical use in aesthetics since its approval by the FDA in 2012, but no rigorous clinical trials have been published to quantify the effect of the skin tightening in any body area. In current clinical practice, the device is frequently used in conjunction with liposuction and both blunt and ultrasound assisted dissection cannulas are utilized. There is some thought that ultrasound assisted dissection may impart some tissue warming and skin tightening effects, but these effects are anecdotal at this time and not rigorously scientifically tested. Our study is designed to address these practice gaps by quantifying the improvement in skin laxity by objective measurements and comparing results obtained between blunt and ultrasound assisted dissection techniques without concurrent liposuction.

This study will use a single-blind, prospective, right-left sided comparator design to assess the effect of the Renuvion/J-Plasma CAP device on skin tightening of upper extremity skin laxity and compare the effect of blunt dissection versus ultrasound assisted site preparation on the procedure results in a non-inferiority design. This study will be a prospective, single-blind (assessor), randomized right-left sided, non-inferiority clinical trial.

Procedures:

This is a randomized, right-left arm, single blinded, prospective noninferiority clinical trial comparing ultrasound assisted to traditional blunt dissection in site preparation prior to subdermal application of the Renuvion/J-plasma cold atmospheric plasma (CAP) device while quantitatively evaluating the efficacy of the Renuvion device.

A total of 15 patients will be enrolled. Dropout is anticipated to be low as the study visits will concur with routine clinical follow up appointments. The number needed to treat to show noninferiority between blunt dissection and ultrasound assisted dissection is 13 and the number needed to treat to show statistically significant difference between baseline and follow up is 3 for the Renuvion/J-Plasma procedure.

DETAILED DESCRIPTION:
The Renuvion/J-plasma cold atmospheric plasma device has been in clinical use in aesthetics since its approval by the FDA in 2012, but no rigorous clinical trials have been published to quantify the effect of the skin tightening in any body area. In current clinical practice, the device is frequently used in conjunction with liposuction and both blunt and ultrasound assisted dissection cannulas are utilized. There is some thought that ultrasound assisted dissection may impart some tissue warming and skin tightening effects, but these effects are anecdotal at this time and not rigorously scientifically tested. Our study is designed to address these practice gaps by quantifying the improvement in skin laxity by objective measurements and comparing results obtained between blunt and ultrasound assisted dissection techniques without concurrent liposuction.

Study Design:

This study will use a single-blind, prospective, right-left sided comparator design to assess the effect of the Renuvion/J-Plasma CAP device on skin tightening of upper extremity skin laxity and compare the effect of blunt dissection versus ultrasound assisted site preparation on the procedure results in a non-inferiority design. This study will be a prospective, single-blind (assessor), randomized right-left sided, non-inferiority clinical trial.

Bliniding:

To blind the study, the sub-investigator/operator will use an internet-based random number generator to assign the right arm to blunt dissection (odd numbers) or ultrasound-assisted dissection (zero and even numbers). Due to the nature of the procedure, it will be impossible to blind the operator and the patient to site preparation technique. The assessors and coordinators will remain blinded to the treatment assignment throughout the study. Measurements and photographs will not be labeled regarding which site preparation method was used. A patient specific paper chart will have treatment assignments, which will minimize the potential for inadvertent unblinding and allow for unblinding in the event unblinding becomes necessary.

Study Purposes and Objectives:

1. Quantify the clinical improvement from baseline to 1, 3 and 9 months after treatment of underarm laxity using the Renuvion/J-Plasma cold atmospheric plasma (CAP) device with both Vaser ultrasound-assisted dissection and blunt dissection methods for site preparation in a randomized, right-left arm single blinded, prospective clinical trial.

   1. Compare ultrasound-assisted site prepared side baseline photographs to 1-month, 3-month, and 9-month post-treatment photos to assess change in area between overlaid photographs taken in both sagittal and coronal planes.
   2. Compare ultrasound-assisted site prepared side baseline photographs to 1-month, 3-month, and 9 month post-treatment photos to assess change in distance of lowest hanging point between overlaid photographs taken in both sagittal and coronal planes.
   3. Compare ultrasound-assisted site prepared side linear circumference at baseline to 1-month, 3-month, and 9-month post-treatment measurements to assess change in linear circumference of treated area.
   4. Compare blunt dissection site prepared side baseline photographs to 1-month, 3-month, and 9-month post-treatment photos to assess change in area between overlaid photographs taken in both sagittal and coronal planes.
   5. Compare blunt dissection site prepared side baseline photographs to 1-month, 3-month, and 9-month post-treatment photos to assess change in distance of lowest hanging point between overlaid photographs taken in both sagittal and coronal planes.
   6. Compare blunt dissection site prepared side linear circumference at baseline to 1-month, 3-month, and 9-month post-treatment measurements to assess change in linear circumference of treated area.
2. Compare non-inferiority of clinical endpoints between blunt dissection cannula and Vaser ultrasound-assisted cannula for site preparation of Renuvion/J-Plasma treatment at 1, 3, and 9 months post treatment.

   1. Compare ultrasound-assisted site prepared side to blunt dissection prepared side by calculating the difference in area change in sagittal and coronal planes as determined in objective 1 between the two treatment modalities.
   2. Compare ultrasound-assisted site prepared side to blunt dissection prepared side by calculating the difference in lowest hanging point change in sagittal and coronal planes as determined in objective 1 between the two treatment modalities.
   3. Compare ultrasound-assisted site prepared side to blunt dissection prepared side by calculating the difference in linear circumference of treated area change as determined in objective 1 between the two treatment modalities.
3. Assess patient reported outcomes of the treatment using the BODY-Q and Skindex-16 instruments.

Procedures:

This is a randomized, right-left arm, single blinded, prospective noninferiority clinical trial comparing ultrasound assisted to traditional blunt dissection in site preparation prior to subdermal application of the Renuvion/J-plasma cold atmospheric plasma (CAP) device while quantitatively evaluating the efficacy of the Renuvion device.

A total of 15 patients will be enrolled. Dropout is anticipated to be low as the study visits will concur with routine clinical follow up appointments. The number needed to treat to show noninferiority between blunt dissection and ultrasound assisted dissection is 13 and the number needed to treat to show statistically significant difference between baseline and follow up is 3 for the Renuvion/J-Plasma procedure. The study timeline is summarized in table 1.

Screening:

For screening, subjects with qualifying underarm skin laxity without excess fat will be asked to read and sign the informed consent document. They will be reminded that they are to take their time, and if necessary, take it home for further consideration. Questions will be answered. Those meeting inclusion / exclusion criteria who have signed informed consent will be enrolled.

After answering questions and prior to the treatment, the Principal Investigator (PI) will examine the upper body of the patient and assess the type of upper arm skin laxity, amount of underlying fat, and perform measurements to include weight, mid-biceps arm circumference and skin ptosis from brachial sulcus to the lowermost border of pendulous skin. Standardized photographs of the treatment area will be obtained in sagittal and coronal planes of the arms abducted to 90o with elbows flexed to 90o. The patient will complete the Body-Q and Skindex-16 patient reported outcomes measurement tools.

Using a random number generator, the patient will be randomized to undergo blunt dissection vs ultrasound-assisted dissection of the right arm. The left arm will receive the site preparation modality not selected for the right arm. The sub-investigator will perform the randomization on the day of the procedure and the PI will be blinded to the treatment assignment.

At follow up visits, the blinded PI will perform an upper body exam and repeat mid-biceps arm circumference and skin ptosis measurements. Standardized photographs will be repeated in sagittal and coronal planes as at baseline. The patient will complete the Body-Q and Skindex-16 patient reported outcomes measurement tools. Treatment related adverse event information will be collected.

Adverse events:

Evaluations for adverse events will be carried out by the PI or sub-I at scheduled follow up visits or if the clinic is notified of problems by the patient. If adverse events have not resolved at the time of the final visit, the patient will be followed for resolution of these events by phone or office visits. Specific adverse events to be tracked will include pain, bleeding, hematoma formation, infection, nerve damage, scarring, and skin discoloration in the treatment sites. Major cardiac and neurologic events will also be noted, but are not anticipated based on existing data on these and similar procedures.

Procedure:

The patient will arrive on the day of the procedure and sites will be prepped in a standard sterile fashion. Patients will receive diazepam and midazolam orally as appropriate for anxiolysis or mild sedation. Local anesthesia will be administered using tumescent lidocaine (1 g lidocaine and 1 mg epinephrine in 100 ml plus 10 mEq sodium bicarbonate in 10 ml added to 1000 ml of 0.9% physiologic saline) at a maximum dose of 28 mg/kg to prevent toxicity. 4 mm incisions will be made at the distal portion of the posterior upper arm, approximately 2.5-4 cm from the olecranon process when the arm is at 90 degrees of flexion, and at the most proximal portion of the posterior upper arm in the axillary crease. A standard 3 mm blunt liposuction cannula not attached to suction will be used to dissect the subcutaneous tissue of the posterior upper arm on the side randomized to blunt dissection. Several passes will be made using the blunt dissection cannula with (increasing/decreasing sizes) until the dissection plane has been completed. The Renuvion/J-Plasma CAP device will be inserted into the openings created for the dissection and 4 passes of the device applied to the underside of the dermis will be made at a setting of 80mJ and 2.0 L of flow. This process will be repeated on the contralateral side using the ultrasound assisted device (Vaser) in place of the blunt dissection cannula at the setting of 60% energy (10W) for no greater than 2.5 min.

Post-procedure, the cannula wounds will be closed with one 4-0 nylon suture, and otherwise left open to allow for drainage and venting. The upper arms will be wrapped with absorbent pads and an industry standard upper arm compression garment which we will provide. The compression garment is to be worn for 2 weeks following the procedure. Post-operative pain will be managed with acetaminophen and 5mg/325mg hydrocodone/acetaminophen as needed. The patient will shower normally the following day and expect some mild serosanginous drainage from the incision sites over 48 hours following the procedure. After 48 hours the patient will then begin daily placement of a thin layer of white petrolatum over the incision sites followed by a small bandage or Band-aid

Evaluations:

Efficacy evaluations will be performed at baseline, 1-month post-procedure, 3-months post-procedure, and 9-months post-procedure. For each evaluation, a coordinator who is blinded to the treatment assignment will measure upper arm circumference of each arm at the point of maximum diameter and vertical distance from the brachial sulcus to the lowermost border of pendulous skin when the arms are positioned at 90o abducted at the shoulder and 90o flexed at the elbow. Circumference will be measured with a flexible measuring tape and vertical distance will be measured using a rigid ruler. These measurements will be entered into a spreadsheet (Microsoft Excel, Microsoft Corporation, Redmond, WA) and analyzed using R statistical software (R Foundation for Statistical Computing, Vienna, Austria) to determine the mean change from baseline and standard deviation at 1, 3, and 9-months post-procedure and between 1- and 3-months post-procedure, 1- and 9- months post-procedure, and 3- and 9-months post-procedure. T-testing will be performed using the R statistical software package to compare before and after measurements at each time point from baseline and between each follow up interval. P-values will be calculated with a significance level of P < 0.05 being considered significant.

Standardized photographs of the treatment area will be obtained by trained staff photographers in sagittal and coronal planes of the arms abducted to 90o with elbows flexed to 90o. Digital photographs will be obtained at baseline, 1-month post-procedure, 3-months post-procedure, and 9-months post-procedure. Photographs will be obtained using a Canon camera for sagittal, coronal, and oblique views and Visia system (Canfield Scientific, Inc., Parsippany, NJ) for sagittal and oblique views.

The patient will complete the clinically validated Body-Q patient reported outcomes measurement tool for upper arms at baseline, 1, 3, and 9-months post-procedure. A copy of this assessment tool is included in the supporting documents section.

1. Primary Efficacy Measures:

   The efficacy will be measured using the change in area and vertical distance calculated from standardized digital photographic overlays using the sagittal view between baseline and 9-months post-procedure.
2. Secondary Efficacy Measures:

   Unless otherwise stated, secondary efficacy measures will be calculated between baseline and 1-month post-procedure, baseline and 3-months post-procedure, baseline and 9-months post-procedure, between 1- and 3-months post-procedure, between 1- and 9-months post-procedure, and between 3- and 9-months post-procedure. These measures will include the change in area and vertical distance calculated from standardized digital photographic overlays using the sagittal view for non-primary endpoint time intervals, the change in area and vertical distance calculated from standardized digital photographic overlays using the coronal view, the difference in arm circumference, the difference in measured vertical pendulous skin, and differences in Body-Q and Skindex-16 patient recorded outcomes measurements, and subjective blinded assessor assessments.
3. Adverse events:

Adverse events will be catalogued, detailed, and presented in table format.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to give informed written consent
* BMI < 25
* Age of at least 18 and not greater than 75 years old
* Male or Female
* Ability to undergo procedure
* Stable weight for 6 months
* 2 cm to 6 cm of upper arm ptosis
* Less than or equal to 1 cm of skin pinch thickness in area to be treated.

Exclusion Criteria:

* Prior liposuction to the proposed treatment areas
* Connective tissue disease
* History of Keloidal scarring
* Nursing/pregnant
* Using systemic steroids or immunosuppressants
* Current smoking
* Body dysmorphic disorder
* Allergy or intolerance to tumescent anesthesia
* Prior significant trauma or scarring to the upper arms
* Lymphedema of the upper extremities
* Significant asymmetry in diameter or laxity of upper arms

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Change in baseline area compared to 9 months post procedure from digital photographs. | 9 months
  The efficacy will be measured using the change in area calculated from standardized digital photographic overlays using the sagittal view between baseline and 9-months post-procedure.
Change in vertical distance compared to 9 months post procedure from digital photographs | 9 months
  The efficacy will be measured using the change in vertical distance calculated from standardized digital photographic overlays using the sagittal view between baseline and 9-months post-procedure.

SECONDARY OUTCOMES:
Change in baseline area compared to 1 months post procedure from digital photographs. | 1 month
  This measurement will include the change in area calculated from standardized digital photographic overlays using the sagittal view for non-primary endpoint time intervals, the change in area calculated from standardized digital photographic overlays using the coronal view.
Change in baseline vertical distance compared to 1 months post procedure from digital photographs. | 1 month
  This measurement will include the change in vertical distance calculated from standardized digital photographic overlays using the sagittal view for non-primary endpoint time intervals, the change in area calculated from standardized digital photographic overlays using the coronal view.
Change in baseline area compared to 3 months post procedure from digital photographs. | 3 months
  This measurement will include the change in area calculated from standardized digital photographic overlays using the sagittal view for non-primary endpoint time intervals, the change in area calculated from standardized digital photographic overlays using the coronal view.
Change in vertical distance compared to 3 months post procedure from digital photographs. | 3 months
  This measurement will include the change in vertical distancecalculated from standardized digital photographic overlays using the sagittal view for non-primary endpoint time intervals, the change in area calculated from standardized digital photographic overlays using the coronal view.
Change in arm circumference from baseline to 9 months. | 9 months
  Change in arm circumference from baseline to 9 months.
Change in Body-Q scores from baseline to 9 months | 9 months
  The BODY-Q includes 13 appearance scales that measure satisfaction with the body overall and specific parts of the body in terms of size, shape, dressed, naked, in photos, etc. The BODY-Q includes 10 quality of life scales. For screening purposes, the BODY-Q has scales that measure expectations on how appearance and quality of life might change after treatment and appearance-related distress. The BODY-Q measures important outcomes in weight loss and body contouring, including body image and physical, social, psychological and sexual function. The BODY-Q has a set of 4 scales that can be used as quality metrics. These scales measure satisfaction with information provided (about complications, healing and recovery time and details of the procedure) as well as the surgeon, medical team and office staff.
Change in Skindex-16 scores from baseline to 9 months | 9 months
  The Skindex-16 is a validated questionnaire that uses an analog scale from 0 (best) to 6 (worst) to measure emotional and functional symptoms related to the skin. Skindex accurately and sensitively measures how much patients are bothered by their skin conditions.

CONTACTS AND LOCATIONS:
Overall Officials: David Smart, M.D., Principal Investigator — University of Utah MidValley Dermatology
Locations (1):
- University of Utah MidValley Dermatology, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wong R, Geyer S, Weninger W, Guimberteau JC, Wong JK. The dynamic anatomy and patterning of skin. Exp Dermatol. 2016 Feb;25(2):92-8. doi: 10.1111/exd.12832. Epub 2015 Oct 13. PMID 26284579
- [Result] Gutowski KA. Microfocused Ultrasound for Skin Tightening. Clin Plast Surg. 2016 Jul;43(3):577-82. doi: 10.1016/j.cps.2016.03.012. Epub 2016 May 4. PMID 27363772
- [Result] Gentile RD. Renuvion/J-Plasma for Subdermal Skin Tightening Facial Contouring and Skin Rejuvenation of the Face and Neck. Facial Plast Surg Clin North Am. 2019 Aug;27(3):273-290. doi: 10.1016/j.fsc.2019.03.001. Epub 2019 May 22. PMID 31280843
- [Result] Fakhouri TM, El Tal AK, Abrou AE, Mehregan DA, Barone F. Laser-assisted lipolysis: a review. Dermatol Surg. 2012 Feb;38(2):155-69. doi: 10.1111/j.1524-4725.2011.02168.x. Epub 2011 Oct 20. PMID 22093156
- [Result] Dong J, Amir Y, Goldenberg G. Advances in minimally invasive and noninvasive treatments for submental fat. Cutis. 2017 Jan;99(1):20-23. PMID 28207010